CLINICAL TRIAL: NCT02642614
Title: A Phase I Randomized, Double-blind, Placebo-controlled, Parallel-group Trial of BI 1026706 Administered Orally as Tablets Twice Daily for 4 Weeks to Patients With COPD in Order to Evaluate Safety, Tolerability, Pharmacokinetics and Effect on Inflammation
Brief Title: Safety, Tolerability and Pharmacokinetics and Effect on Inflammation of Oral BI 1026706 in Patients With COPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1320.16; 2015-002123-25 (EudraCT Number)
Record Dates: First submitted 2015-12-23; First posted 2015-12-30 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- BI 1026706 low dose (Experimental)
  Interventions: Drug: BI 1026706; Drug: Placebo
- BI 1026706 medium (Experimental)
  Interventions: Drug: BI 1026706; Drug: Placebo
- BI 1026706 high dose (Experimental)
  Interventions: Drug: BI 1026706; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1026706
  Arms: BI 1026706 high dose; BI 1026706 low dose; BI 1026706 medium
Drug: Placebo
  Arms: Placebo
Drug: Placebo — For blinding purposes

SUMMARY:
The main objective of the current trial is to investigate safety, tolerability, pharmacokinetics and effect on inflammation of oral BI 1026706 administered twice daily for 4 weeks in patients with COPD.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent consistent with ICH-Good Clinical Practice (GCP) guidelines and local legislation prior to participation in the trial. Medication washout and medication restrictions are allowed only after signed informed consent is obtained.
* Males or females not of childbearing potential between 40 and 80 years (each inclusive) of age, on the day of patient´s signature of informed consent.
* All patients must have a documented diagnosis of COPD according to Global Initiative for Chronic Obstructive Lung Disease (GOLD).
* Post-bronchodilator forced expiratory volume (FEV)1 of >=40% and <=90% of predicted normal at Visit 1
* Post-bronchodilator FEV1/forced vital capacity (FVC) <70% at Visit 1
* Patients must be current or ex-smokers with a smoking history of more than 10 pack years
* Patients on stable respiratory medications for at least 6 weeks prior to randomization (Visit 3).
* Patients must be able to perform technically acceptable pulmonary function tests.

Exclusion criteria:

* Significant pulmonary disease other than COPD or other medical conditions as determined by medical history, examination, and clinical investigations at screening that may, in the opinion of the investigator, result in the any of the following:

  1. Put the patient at risk because of participation in the study
  2. Influence the results of the study
  3. Cast doubt on the patients ability to participate in the study
* Patients with current asthma. For patients with allergic rhinitis or atopy, source documentation is required to verify that the patient does not have asthma.
* Patients with clinically relevant abnormal hematology, blood chemistry, or urinalysis at the screening visit (Visit 1), if the abnormality indicates a relevant disease as defined in exclusion criterion number 1. Safety laboratory screening evaluation (Visit 1) can be repeated a maximum of two times.
* Patients with a history of myocardial infarction or apoplexy within 6 months of the screening visit (Visit 1) or between the screening visit (Visit 1) and randomization.
* Patients with a history of and/or active life-threatening cardiac arrhythmia, as assessed by the investigator.
* Patients with a marked baseline prolongation of QT/QTcB interval (such as repeated demonstration of a QTcB interval >450 ms), pulse/heart rate outside 50 to 90 bpm at Visit 1 (if confirmed by pulse rate measurement over 60 seconds), or any other relevant ECG finding.
* Patients with a history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome).
* Patients with known active tuberculosis.
* Patients with clinically relevant bronchiectasis, as assessed by the investigator.
* Patients with any respiratory infection (such as common cold, acute sinusitis, or similar illnesses) or COPD exacerbation within 6 weeks prior to the screening visit (Visit 1) or between the screening visit and randomization.
* Patients who have undergone thoracotomy with pulmonary resection (patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1).
* Patients with a malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last 5 years. Patients with treated basal cell carcinoma or fully cured squamous cell carcinoma are allowed to participate.
* Patients with a history of and/or active significant alcohol or drug abuse as assessed by the investigator.
* Patients who are being treated with non-permitted concomitant medication.
* Patients who have taken an investigational drug within 4 weeks prior to Visit 1 or if screening occurs within six half-lives of intake of another investigational drug (whichever is greater).
* Patients with surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication as assessed by the investigator.
* Patients with veins unsuited for venipuncture (for instance, veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture) as assessed by the investigator.
* Patients who are unable to comply with the dietary regimen.
* Patients who have been previously randomized in this study.
* Patients who have donated more than 100 mL blood in the 4 weeks prior to Visit 1 and between Visit 1 and Visit 3 or patients who have the intention to donate blood between Visit 3 and four weeks after the end of trial visit.
* Patients who are pregnant or breastfeeding
* Male patients who do not agree to minimize the risk of female partners becoming pregnant from the first dosing day until 3 months after the trial medication treatment has finished.
* Patient is assessed as unsuitable for inclusion by the investigator; for instance, because he or she is not considered to comply with study requirements

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2016-06-14 (Actual); Study Completion 2016-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (10):
- Denmark (2):
  - Bispebjerg og Frederiksberg Hospital, København NV
  - Odense University Hospital, Odense C
- Germany (6):
  - PAREXEL International GmbH, Berlin
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Inamed GmbH, Gauting
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Fraunhofer ITEM, Hanover
  - KLB Gesundheitsforschung Lübeck GmbH, Lübeck
- Skånes universitetssjukhus, Lund, Lund, Sweden
- The Medicines Evaluation Unit, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Double dummy trial, 2 different type of medication were dispensed to the patient with the help of two different bottles: Bottle 1 - 5 mg OR 25 mg BI 1026706 tablets or placebo tablets matching 5 mg and 25 mg BI 1026706 tablets, Bottle 2 -100 mg tablets or Placebo tablets matching 100 mg BI 1026706 tablets.
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be entered in to the trial if any of the specific entry criteria was violated.
Groups:
- Placebo: Patients received one placebo tablet (twice daily (BID) matching the 5 and 25 milligram (mg) tablets and one placebo tablet matching the 100 mg tablet orally with water with or without food (except on the morning of Days 1 and 28 when patients were to fast overnight for at least 8 hours before administration of trial medication) for 28 days, with end-of-trial visit 5 to 10 days after last administration of trial medication. In the twice daily (BID) dosing regimen, the patient had to take 2 tablets in the morning and 2 tablets in the evening.
- 5 Milligram BI 1026706: Patients received BI 1026706 (5 milligram (mg) twice daily (BID) along with placebo matching the 100 mg tablet) film-coated tablet administered orally with water with or without food (except on the morning of Days 1 and 28 when patients were to fast overnight for at least 8 hours before administration of trial medication) for 28 days, with end-of-trial visit 5 to 10 days after last administration of trial medication.
- 25 Milligram BI 1026706: Patients received BI 1026706 (25 milligram (mg) twice daily (BID) along with placebo matching the 100 mg tablet) film-coated tablet administered orally with water with or without food (except on the morning of Days 1 and 28 when patients were to fast overnight for at least 8 hours before administration of trial medication) for 28 days, with end-of-trial visit 5 to 10 days after last administration of trial medication.
- 100 Milligram BI 1026706: Patients received BI 1026706 (100 milligram (mg) twice daily (BID) along with placebo matching the 5 and 25 mg tablets) film-coated tablet administered orally with water with or without food (except on the morning of Days 1 and 28 when patients were to fast overnight for at least 8 hours before administration of trial medication) for 28 days, with end-of-trial visit 5 to 10 days after last administration of trial medication.
Period: Overall Study
Arm/Group | Placebo | 5 Milligram BI 1026706 | 25 Milligram BI 1026706 | 100 Milligram BI 1026706
Started | 30 | 30 | 30 | 30
Completed | 27 | 28 | 28 | 28
Not Completed | 3 | 2 | 2 | 2
Not completed — Adverse Event | 1 | 1 | 2 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set (RS): The RS included all patients who were randomized, whether treated or not. The treatment assignment was determined based on the treatment arm to which the patient was randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 5 Milligram BI 1026706 | 25 Milligram BI 1026706 | 100 Milligram BI 1026706 | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (8.5) | 65.7 (7.2) | 65.3 (6.1) | 62.5 (7.1) | 64.3 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 11 | 10 | 41
  Male | 19 | 21 | 19 | 20 | 79

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of BI 1026706, as Assessed by Frequency (in Percent) of Patients With Treatment Emergent Adverse Events (TEAEs) Over the Treatment Period.
Description: Safety and tolerability of BI 1026706, as assessed by frequency (in percent) of patients with treatment-emergent adverse events (TEAEs) over the treatment period.
Time Frame: From first drug administration until 4 days after last drug administration, up to 32 days
Population: Treated set (TS): The TS included all patients who were randomized and treated with at least 1 dose of trial medication. The treatment assignment was determined based on the first treatment the patient received.
Measure: Number; unit: Percentage of Patients
Arm/Group | Placebo | 5 Milligram BI 1026706 | 25 Milligram BI 1026706 | 100 Milligram BI 1026706
Number analyzed (Participants) | 30 | 30 | 30 | 30
Percentage of Patients | 60.0 | 46.7 | 66.7 | 53.3

2. Secondary Outcome: Change in Absolute Number of Neutrophil in Sputum at the End of the Planned Treatment Period
Description: Change in Absolute Number of Neutrophil in Sputum at the end of the planned treatment period
Time Frame: 28 days
Population: Treated set including participants with available data for the endpoint percent change in absolute number of neutrophil in sputum at the end of the planned treatment period
Measure: Mean (Standard Error); unit: 10^6 cells/ milliliter (mL)
Arm/Group | Placebo | 5 Milligram BI 1026706 | 25 Milligram BI 1026706 | 100 Milligram BI 1026706
Number analyzed (Participants) | 23 | 22 | 25 | 25
10^6 cells/ milliliter (mL) | 2.12 (0.47) | 3.37 (0.79) | 3.35 (0.73) | 3.06 (0.66)
Statistical Analysis 1: Comparison: Placebo vs 5 Milligram BI 1026706; Adjusted means were calculated by exponentiating Least Square (LS) means of corresponding values obtained from fitting an ANCOVA model to the natural log transformed endpoint variable, including treatment effect and study baseline as covariates, and adjusting for stratification factors (extensive pharmacokinetic (PK) sub-study participation and Multiple-breath washout (MBW) sub-study participation); Test type: Superiority or Other; p = 0.1540, ANCOVA; Ratio of adjusted mean = 1.59, 90% CI 2-sided [0.93 to 2.72], Standard Error of Mean 0.51 — Standard Error of Mean is actually "Standard Error of ratio of adjusted means", adjusted means ratio is calculated as 5 milligram BI 1026706 divided by Placebo
Statistical Analysis 2: Comparison: Placebo vs 25 Milligram BI 1026706; The adjusted means were calculated by exponentiating the LS means of the corresponding values obtained from fitting an ANCOVA model to the natural log transformed endpoint variable, including treatment effect and study baseline as covariates, and adjusting for stratification factors (extensive PK sub-study participation and MBW sub-study participation); Test type: Superiority or Other; p = 0.1430, ANCOVA; Ratio of adjusted mean = 1.58, 90% CI 2-sided [0.94 to 2.65], Standard Error of Mean 0.49 — Standard Error of Mean is actually "Standard Error of ratio of adjusted means", adjusted means ratio is calculated as 25 milligram BI 1026706 divided by Placebo
Statistical Analysis 3: Comparison: Placebo vs 100 Milligram BI 1026706; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.2398, ANCOVA; Ratio of adjusted mean = 1.44, 90% CI 2-sided [0.86 to 2.41], Standard Error of Mean 0.45 — Standard Error of Mean is actually "Standard Error of ratio of adjusted means", adjusted means ratio is calculated as 100 milligram BI 1026706 divided by Placebo

3. Secondary Outcome: Maximum Measured Concentration of BI 1026706 in Plasma (Cmax) After the First Dose (Morning of Day 1)
Description: Maximum measured concentration of BI 1026706 in plasma (Cmax) after the first dose (morning of Day 1)
Time Frame: -0:10 hour(h) before drug administration and 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, and 12:00h after drug administration.
Population: Extensive pharmacokinetic set (ePKS): The ePKS included all patients in the PKS who signed the informed consent for participating in the extensive PK sub-study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles (nmol) / litre (L)
Arm/Group | 5 Milligram BI 1026706 | 25 Milligram BI 1026706 | 100 Milligram BI 1026706
Number analyzed (Participants) | 10 | 11 | 11
nanomoles (nmol) / litre (L) | 39.0 (47.7) | 145 (37.8) | 524 (39.0)

4. Secondary Outcome: Time From Dosing to Maximum Concentration of BI 1026706 in Plasma (Tmax) After the First Dose (Morning of Day 1)
Description: Time from dosing to maximum concentration of BI 1026706 in plasma (Tmax) after the first dose (morning of Day 1)
Time Frame: as for outcome 3
Population: ePKS
Measure: Median (Full Range); unit: hour
Arm/Group | 5 Milligram BI 1026706 | 25 Milligram BI 1026706 | 100 Milligram BI 1026706
Number analyzed (Participants) | 10 | 11 | 11
hour | 1.00 (47.7) [0.500 to 2.00] | 1.02 (37.8) [0.500 to 3.00] | 1.00 (39.0) [0.483 to 3.00]

5. Secondary Outcome: Area Under the Concentration-time Curve of BI 1026706 in Plasma (AUC 0-12h) After the First Dose (Morning of Day 1)
Description: Area under the concentration-time curve of BI 1026706 in plasma (AUC 0-12h) after the first dose (morning of Day 1)
Time Frame: as for outcome 3
Population: ePKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles (nmol) * hour (h) / litre (L)
Arm/Group | 5 Milligram BI 1026706 | 25 Milligram BI 1026706 | 100 Milligram BI 1026706
Number analyzed (Participants) | 10 | 11 | 11
nanomoles (nmol) * hour (h) / litre (L) | 138 (58.2) [0.500 to 2.00] | 489 (44.4) [0.500 to 3.00] | 1840 (42.7) [0.483 to 3.00]

6. Secondary Outcome: Maximum Measured Concentration of BI 1026706 in Plasma at Steady State Over a Uniform Dosing Interval Tau (Cmax, ss) After the Last Dose (Morning of Day 28)
Description: Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval tau (Cmax, ss) after the last dose (morning of Day 28)
Time Frame: as for outcome 3
Population: ePKS including participants with available data for this endpoint
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 5 Milligram BI 1026706 | 25 Milligram BI 1026706 | 100 Milligram BI 1026706
Number analyzed (Participants) | 9 | 9 | 10
nmol/L | 51.2 (26.4) [0.500 to 2.00] | 185 (34.7) [0.500 to 3.00] | 870 (37.9) [0.483 to 3.00]

7. Secondary Outcome: Time From Dosing to Maximum Concentration of BI 1026706 in Plasma (Tmax, ss) After the Last Dose (Morning of Day 28)
Description: Time from dosing to maximum concentration of BI 1026706 in plasma (Tmax, ss) after the last dose (morning of Day 28)
Time Frame: as for outcome 3
Population: ePKS including participants with available data for this endpoint
Measure: Median (Full Range); unit: hour
Arm/Group | 5 Milligram BI 1026706 | 25 Milligram BI 1026706 | 100 Milligram BI 1026706
Number analyzed (Participants) | 9 | 9 | 10
hour | 1.00 (26.4) [0.500 to 3.00] | 1.50 (34.7) [1.00 to 3.00] | 0.767 (37.9) [0.500 to 3.00]

8. Secondary Outcome: Area Under the Concentration-time Curve of BI 1026706 in Plasma at Steady State Over a Uniform Dosing Interval Tau (AUC Tau, ss) After the Last Dose (Morning of Day 28)
Description: Area under the concentration-time curve of BI 1026706 in plasma at steady state over a uniform dosing interval tau (AUC tau, ss) after the last dose (morning of Day 28)
Time Frame: as for outcome 3
Population: ePKS including participants with available data for this endpoint
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 5 Milligram BI 1026706 | 25 Milligram BI 1026706 | 100 Milligram BI 1026706
Number analyzed (Participants) | 9 | 9 | 10
nmol*h/L | 197 (47.1) [0.500 to 3.00] | 781 (40.7) [1.00 to 3.00] | 3850 (34.3) [0.500 to 3.00]

ADVERSE EVENTS:
Time Frame: From first drug administration until 4 days after last drug administration, up to 32 days
Arm/Group | Placebo | 5 Milligram BI 1026706 | 25 Milligram BI 1026706 | 100 Milligram BI 1026706
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/30 | 2/30 | 0/30
Other Adverse Events (participants affected / at risk) | 16/30 | 12/30 | 13/30 | 10/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | 5 Milligram BI 1026706 (N=30) | 25 Milligram BI 1026706 (N=30) | 100 Milligram BI 1026706 (N=30)
Visual field defect (Nervous system disorders) | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | 5 Milligram BI 1026706 (N=30) | 25 Milligram BI 1026706 (N=30) | 100 Milligram BI 1026706 (N=30)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 4 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1 | 3
Oral herpes (Infections and infestations) | 2 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 3 | 3 | 3 | 3
Forced expiratory volume decreased (Investigations) | 8 | 8 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Headache (Nervous system disorders) | 4 | 0 | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.